CLINICAL TRIAL: NCT01623661
Title: Effect of Intravenous Sodium Chloride on Urinary Biomarkers for Measurement of Sodium- and Water Channel Activity in the Nephron in Healthy Subject an Patients With Chronic Kidney Disease. A Case Control Study
Brief Title: Effect of Hypertonic Sodium Chloride on Urinary Biomarkers in Healthy Subjects and Patients With Chronic Kidney Disease
Acronym: CASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, DMSc, Regional Hospital Holstebro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EBP-JMJ-2012-2
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Nephropathy
Keywords: Nephrology; chronic kidney disease; sodium-channels; water-channels; BCM
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hypertonic saline (Other): hypertonic saline 3.0% (7 ml/kg)
  Interventions: Other: hypertonic saline

INTERVENTIONS:
Other: hypertonic saline — hypertonic saline 3.0 % (7 ml/kg)
  Other Names: hypertonic NaCl

SUMMARY:
Patients with chronic kidney disease (CKD) have a defect in the tubular reabsorption of sodium, and therefore the ability to excrete a sodium load is diminished compared to healthy subjects.

Urinary biomarkers reflects the water- and sodium-channel activity in the kidney and may be measured after an infusion with hypertonic saline in CKD patients and healthy subjects.

DETAILED DESCRIPTION:
The fractional sodium excretion is elevated as high as 10-20% In patients with chronic kidney disease (CKD) Changes in the sodium intake results in a slower expansion and/or reduction in extracellular fluid in CKD patients.

Urinary biomarkers reflects the kidneys transport of sodium and water in the nephron.

Changes in the sodium-and water channel activity is induced by intervention with hypertonic Saline (3.0%) The change in sodium-and water channel activity is followed by change in extracellular and intracellular fluid compartments and the plasma concentration of vasoactive hormones.

The purpose of this study is to investigate the changes in urinary biomarkers (u-NKCC2, u-ENaC-gamma and u-AQP2), the activity of the sodium-and water channels, the extra- and intracellular fluid compartments and the plasma concentration of Vasoactive hormones in patients with CKD and in healthy subjects.

Subjects and patients are examined during one examination day. Four days prior to the examination day the subjects consume a standardized diet based on the amount of sodium and calories. On the examination day the subjects receive an infusion with hypertonic saline.

Renal function is measured by renal clearance of 51Cr-EDTA. Urinary biomarkers (u-NKCC2, u-ENaC-gamma and u-AQP2) are measured to evaluate the activity of sodium channels in the nephron and changes in fluid compartments are measured by body composition monitor.

ELIGIBILITY:
Inclusion Criteria:

1. healthy subjects

   * healthy males and females
   * age 18-70
   * BMI range 18,5-30,0 kg/m2
2. Patients with CKD

   * age 18-70
   * eGFR 15-60 ml/min
   * BMI range 18.5 - 30.0 kg/m2

Exclusion Criteria:

1. healthy subjects

   * hypertension (ie ambulatory BP >130 mmHg systolic or/and >80 mmHg diastolic)
   * history or clinical significant signs of heart, lung, liver, kidney, endocrine, brain or neoplastic disease.
   * alcohol abuse
   * drug abuse
   * smoking
   * pregnancy or nursing
   * blood donation within a month prior to examination
   * Medical treatment apart from oral contraception
2. Patients with chronic kidney disease

   * clinical significant signs of heart, lung, liver, endocrine, brain or neoplastic disease.
   * diabetes
   * immunosuppressive medications
   * smoking
   * alcohol abuse
   * drug abuse
   * pregnancy or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
urinary biomarkers | one day
  Urinary epithelial sodium channels (ENaC), Sodium-potassium-2chloride transporters (NKCC) and aquaporin2 channels (AQP2) before, during and after fluid infusion

SECONDARY OUTCOMES:
vaso active hormones | one day
  plasma concentrations of: renin, Angiotensin II, aldosterone, Vasopressin, atrial natriuretic peptide (ANP) and brain natriuretic peptide (BNP)
extra-and intracellular volume | 6 hours
  measured by body composition monitor at baseline and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, DMSc, Study Director — Regional Hospital Holstebro
Locations (1):
- Medical Research, Holstebro, Denmark

REFERENCES:
- [Derived] Jensen JM, Mose FH, Kulik AE, Bech JN, Fenton RA, Pedersen EB. Abnormal urinary excretion of NKCC2 and AQP2 in response to hypertonic saline in chronic kidney disease: an intervention study in patients with chronic kidney disease and healthy controls. BMC Nephrol. 2014 Jun 26;15:101. doi: 10.1186/1471-2369-15-101. PMID 24970686